CLINICAL TRIAL: NCT02567812
Title: Prospective Data Collection of Patients With Pelvic Inflammatory Disease
Brief Title: Database of Pelvic Inflammatory Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, Kangbuk Samsung Hospital
Other Study IDs: 2015-04-009
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Inflammatory Pelvic Disease
MeSH Terms: conditions — Pelvic Inflammatory Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- In-patient with PID: In-patient with PID who diagnosed at Kangbuk Samsung Hospital

SUMMARY:
The aim of this prospective study is to collect data on in-patients with pelvic inflammatory disease(PID) at Kangbuk Samsung Hospital.

DETAILED DESCRIPTION:
The aim of this prospective study is to collect data on in-patients with pelvic inflammatory disease(PID) at Kangbuk Samsung Hospital. If patients agree to participate in this clinical trial, patient's data (such as age, body mass index, preoperative findings, laboratory findings, radiologic findings, operative findings, pathologic findings, postoperative findings) will be collected in a research database. The research database will be updated, every 6 month, to include data on patient's disease outcome and follow-up care. Although most data will be collected form the medical record, patient may agin be contacted so that researchers can collection some data if it is not in the medical record.

ELIGIBILITY:
Inclusion Criteria:

* All in-patient with PID who diagnosed at Kangbuk Samsung Hospital

Exclusion Criteria:

* Secondary PID caused by other surgical problem or disease
* An inability to fill-up the informed consent

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pelvic inflammatory disease or pelvic inflammatory disorder (PID) is an infection of the upper part of the female reproductive system namely the uterus, fallopian tubes, or the ovaries. Often there may be no symptoms. Signs and symptoms, when present may include lower abdominal pain, vaginal discharge, fever, burning with urination, pain with sex, or irregular menstruation. Untreated PID can result in long term complications including infertility, ectopic pregnancy, chronic pelvic pain, and cancer.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-10; Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
PID database | 10 years
  number of participants with pelvic inflammatory disease

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD PhD, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea